CLINICAL TRIAL: NCT00955630
Title: Intravitreal Ranibizumab for the Treatment of Choroidal Neovascularization in Ocular Histoplasmosis Syndrome
Acronym: IVL for OHS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Retina Associates of Kentucky (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Dr. John Kitchens, Md/Principal Investigator, Retina Associates of Kentucky
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF 4147S
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-08

CONDITIONS: Ocular Histoplasmosis Syndrome
Keywords: Histoplasmosis; Lucentis; Ranibizumab; OHS
MeSH Terms: conditions — Histoplasmosis | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monthly injections (Active Comparator): 3 monthly injections of ranibizumab followed by prn injections
  Interventions: Drug: ranibizumab
- PRN injections (Active Comparator): injections of ranibizumab on a prn basis from the start of the study
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — 3 monthly injections of ranibizumab followed by prn injections for the remainder of the study
  Other Names: Lucentis
  Arms: Monthly injections
Drug: ranibizumab — prn injections of ranibizumab throughout the study
  Other Names: Lucentis
  Arms: PRN injections

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of intravitreal ranibizumab (Lucentis) in patients with fluid and blood leakage in their eyes due to ocular histoplasmosis.

DETAILED DESCRIPTION:
Patients will be evaluated monthly for one year.

Participants will be assigned to one of two groups:

Group A will receive 3 monthly injections of ranibizumab followed by an as needed injection throughout the remainder of the study Group B will receive injections of ranibizumab on an as needed basis throughout the study

You cannot take part in this study if:

1. You are pregnant or intending to become pregnant in the next 12 months or are nursing an infant
2. You are under the age of 18

ELIGIBILITY:
Inclusion Criteria:

* age 18 or over
* active choroidal neovascularization secondary to ocular histoplasmosis
* Visual acuity between 20/25 and 20/400

Exclusion Criteria:

* pregnancy or intent to become pregnant within the next 12 months
* nursing an infant
* premenopausal women not using contraception
* prior treatment with subfoveal thermal laser
* allergy to sodium fluorescein simultaneous participation in another investigation or trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
incidence and severity of ocular adverse events as identified by eye examination | 1 year
incidence and severity of other adverse events as identified by physical examination, subject reporting, and changes in vital signs | 12 mos

SECONDARY OUTCOMES:
mean change in visual acuity | 1 year
mean change in central foveal thickness and total macular volume as obtained by ocular coherence tomography | 6 and 12 months
change in fluorescein angiographic outcomes | 12 months
mean number of injections | 12 mos

CONTACTS AND LOCATIONS:
Overall Officials: John Kitchens, MD, Principal Investigator — Retina Associates of Kentucky
Locations (1):
- Retina Associates of Kentucky, Lexington, Kentucky, United States